CLINICAL TRIAL: NCT00368472
Title: An Open-Label Extension Phase of the Double-Blind, Placebo-Controlled, Dose-Escalation, Parallel-Group Study of E2007 (Perampanel) as an Adjunctive Therapy in Patients With Refractory Partial Seizures
Brief Title: 4-Year Open-Label Extension Phase of the Parallel-Group Study of E2007 in Patients With Refractory Partial Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-A001-207
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
Keywords: Refractory; Partial; Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perampanel (Experimental): Participants previously receiving placebo/perampanel in the double blind study, were titrated to receive perampanel 2 mg to 12 mg, once daily during the OLE study
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel 2 mg to 12 mg, once daily during the OLE study

SUMMARY:
The purpose of this study is to determine the safety of perampanel given as adjunctive, long-term treatment in patients with refractory partial onset seizures.

DETAILED DESCRIPTION:
This is an Open-Label Extension (OLE) study for patients who completed the E2007-A001-206 (NCT00144690) or the E2007-G000-208 (NCT00416195) double-blind, placebo-controlled, dose-escalation, parallel-group studies.

This study consisted of 3 periods: OLE Titration (12 weeks), OLE Maintenance (424 weeks), and OLE Follow-up (4 weeks). During the OLE Titration Period, participants were titrated to their maximum tolerated dose (MTD) of perampanel, up to a maximum of 12 mg/day. The OLE Maintenance Period began at completion of the OLE Titration Period; participants remained on the dose achieved at the end of the OLE Titration Period unless dose adjustment for tolerability reasons was necessary. Participants who either withdrew from the study prematurely or completed the OLE Maintenance Period returned for a final visit at the end of the 4-week OLE Follow-up Period.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

1. Have completed all scheduled visits up to and including Visit 8 in the E2007-A001-206 (NCT00144690) study or Visit 9 of the E2007-G000-208 (NCT00416195) study.
2. Are reliable and willing to make themselves available for the study period and are able to record seizures and report adverse events themselves or have a caregiver who can record and report the events.
3. Females of childbearing potential must continue practicing a medically acceptable method of contraception (e.g., abstinence, a barrier method plus spermicide, or Intrauterine device (IUD)) and for 8 weeks after the end of the OLE study. Those women using hormonal contraceptives must also continue using an additional approved method of contraception (e.g., a barrier method plus spermicide, or IUD).
4. Are between the ages of 18 and 70 years of age, inclusive.
5. Are at least 40 kg (88 lb) of weight.
6. Are currently being treated with a stable dose of one, or a maximum of three licensed Anti-epileptic drugs (AEDs) and are known to take their medication(s) as directed.

KEY EXCLUSION CRITERIA:

1. Show evidence of clinically significant disease (cardiac, respiratory, gastrointestinal, renal disease, etc.,) that, in the opinion of the Investigator(s), could affect the participant's safety or trial conduct.
2. Show evidence of significant active hepatic disease and/or bilirubin greater than 1.5 mg/dL. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medication(s) will be allowed if they are less than two times the upper limit of normal (ULN).
3. Show evidence of significant active hematological disease. White blood cell (WBC) count cannot be less than or equal to 2500/microL or an absolute neutrophil count less than or equal to 1000/microL.
4. Clinically significant ECG abnormality, including prolonged QTc (defined as greater than or equal to 450 msec).
5. Presence of major active psychiatric disease. Participants taking a stable dose of selective serotonin reuptake inhibitor (SSRI) antidepressant will be allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2006-10; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (12):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Denver, Colorado
  - Bradenton, Florida
  - Melbourne, Florida
  - Atlanta, Georgia
  - Baltimore, Maryland
  - New Hyde Park, New York
  - Columbus, Ohio
  - West Jordan, Utah
  - Burlington, Vermont
- Australia (3):
  - Chatswood, New South Wales
  - Maroochydore, Queensland
  - Woodville, South Australia
- Belgium (4):
  - Edegem
  - Ghent
  - Leuven
  - Tielt
- Czechia (6):
  - Brno
  - Hradec Králové
  - Olomouc
  - Ostrava
  - Prague
  - Rychnov nad Kněžnou
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (2):
  - Kuopio
  - Tampere
- France (3):
  - Lille
  - Montpellier
  - Ramonville-Saint-Agne
- Germany (4):
  - Berlin
  - Göttingen
  - München
  - Ulm
- Riga, Latvia
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Rotterdam, Netherlands
- Valencia, Spain
- Stockholm, Sweden
- Dundee, United Kingdom

REFERENCES:
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920
- [Derived] Rektor I, Krauss GL, Bar M, Biton V, Klapper JA, Vaiciene-Magistris N, Kuba R, Squillacote D, Gee M, Kumar D. Perampanel Study 207: long-term open-label evaluation in patients with epilepsy. Acta Neurol Scand. 2012 Oct;126(4):263-9. doi: 10.1111/ane.12001. Epub 2012 Aug 23. PMID 22913800

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel: Participants previously receiving perampanel/placebo in the double-blind study, were titrated to receive perampanel 2 mg to 12 mg, once daily in the Open-Label Extension (OLE) study.
Period: Overall Study
Arm/Group | Perampanel
Started | 138
Completed | 33
Not Completed | 105
Not completed — Adverse Event | 22
Not completed — Medication non-compliance | 4
Not completed — Protocol Violation | 2
Not completed — Request of Investigator or Sponsor | 3
Not completed — Withdrawal by Subject | 40
Not completed — Diary non-compliance | 1
Not completed — Other | 32
Not completed — Missing Final Disposition Date | 1

BASELINE CHARACTERISTICS:
Population: Analysis of baseline characteristics are based on the Full Intent to Treat (ITT) Analysis Set, defined as participants who received at least 1 dose of open-label perampanel and had valid seizure data during the OLE study.
Arm/Group | Perampanel
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Non-serious Adverse Events (AEs) and Treatment-emergent Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered an investigational product. A SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening (ie, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was as a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). In this study, treatment emergent AEs (defined as an AE (serious or non-serious) that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) were assessed. The data is presented in the safety section of the results.
Time Frame: From date of first dose of perampanel up to 30 days after the last dose of perampanel or up to approximately 8 years
Population: Safety Analysis Set was defined as participants who received at least 1 dose of open-label perampanel and had at least 1 safety assessment after the first dose of perampanel in the OLE study.
Measure: Number; unit: Participants
Arm/Group | Perampanel
Number analyzed (Participants) | 138
Participants
  Treatment-emergent non-serious AEs | 112
  Treatment-emergent SAEs | 33

2. Secondary Outcome: Percent Change in Seizure Frequency Per 28 Days Relative to Pre-Perampanel Baseline
Description: Seizure frequency was derived from information (seizure count and type) recorded in participant diary. The seizure frequency per 28 days was calculated as the number of seizures divided by the number of days in the interval and multiplied by 28. The percent change in 28-day seizure frequency from baseline was assessed for all partial-onset seizures types. For participants who had been assigned to treatment with perampanel (previous treatment), pre-perampanel Baseline referred to the Prerandomization Phase of the Core Double Blind study. For participants who had been assigned to treatment with placebo (previous treatment), pre-perampanel Baseline was computed from all data during the Core Double Blind study (including Prerandomization Phase) prior to treatment with perampanel.
Time Frame: Baseline up to Week 221
Population: The analysis was based on the Full Intent to Treat (ITT) Analysis Set, defined as participants who received at least 1 dose of open-label perampanel and had valid seizure data during the OLE study.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Perampanel
Number analyzed (Participants) | 138
Percent Change | -31.5 [-99.2 to 576.1]

3. Secondary Outcome: Percentage of Participants Who Experienced a 50% or Greater Reduction in Seizure Frequency Per 28 Days Relative to the Pre-perampanel Baseline
Description: Seizure frequency was derived from information (seizure count and type) recorded in participant diary. The percentage of participants who experienced a 50% or greater reduction in seizure frequency per 28 days relative to the pre-perampanel Baseline (responders) was assessed. For participants who had been assigned to treatment with perampanel (previous treatment), pre-perampanel Baseline referred to the Prerandomization Phase of the Core Double Blind study. For participants who had been assigned to treatment with placebo (previous treatment), pre-perampanel Baseline was computed from all data during the Core Double Blind study (including Prerandomization Phase) prior to treatment with perampanel. The data is presented as percent responders.
Time Frame: Baseline up to week 221
Population: as for outcome 2
Measure: Number; unit: Percent responders
Arm/Group | Perampanel
Number analyzed (Participants) | 138
Percent responders | 36.2

ADVERSE EVENTS:
Time Frame: From date of first dose of perampanel up to 30 days after the last dose of perampanel or up to approximately 8 years
Description: Treatment emergent adverse events (TEAEs) (defined as an adverse event that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) were assessed.
Arm/Group | Perampanel
Serious Adverse Events (participants affected / at risk) | 33/138
Other Adverse Events (participants affected / at risk) | 112/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=138)
Fibula fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac arrest (Cardiac disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Convulsion (Nervous system disorders) | 5
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 5
Grand mal convulsion (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Postictal state (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 4
Sudden unexplained death in epilepsy (General disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Ileitis (Gastrointestinal disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=138)
Hypertension (Vascular disorders) | 6
Fatigue (General disorders) | 17
Irritability (General disorders) | 7
Oedema peripheral (General disorders) | 7
Anxiety (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 7
Contusion (Injury, poisoning and procedural complications) | 12
Fall (Injury, poisoning and procedural complications) | 12
Foot fracture (Injury, poisoning and procedural complications) | 4
Head injury (Injury, poisoning and procedural complications) | 5
Procedural pain (Injury, poisoning and procedural complications) | 4
Skin laceration (Injury, poisoning and procedural complications) | 11
Blood creatine phosphokinase increased (Investigations) | 5
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Ataxia (Nervous system disorders) | 7
Balance disorder (Nervous system disorders) | 5
Convulsion (Nervous system disorders) | 13
Dizziness (Nervous system disorders) | 56
Headache (Nervous system disorders) | 25
Paraesthesia (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 26
Tremor (Nervous system disorders) | 7
Diplopia (Eye disorders) | 6
Vertigo (Ear and labyrinth disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Bronchitis (Infections and infestations) | 6
Influenza (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 14
Rhinitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 11
Viral infection (Infections and infestations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other